CLINICAL TRIAL: NCT02547402
Title: An Open-label Exploratory Study of the Pharmacokinetic Interaction of CXA-10 Administered to Steady State With Pravastatin and Vytorin® (Simvastatin and Ezetimibe) in Healthy Males
Brief Title: A Study of the PK Interaction of CXA-10 With Pravastatin and Vytorin® in Healthy Males
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Complexa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXA-10-203
Record Dates: First submitted 2015-09-02; First posted 2015-09-11 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — CXA-10; Pravastatin; Ezetimibe, Simvastatin Drug Combination; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CXA-10 (Experimental): CXA-10 (10-nitro-9(E)-octadec-9-enoic acid) is a specific isomer of nitrated oleic acid
  Interventions: Drug: CXA-10; Drug: pravastatin; Drug: Vytorin® (combination of simvastatin and ezetimibe)

INTERVENTIONS:
Drug: CXA-10 — CXA-10 (10-nitro-9(E)-octadec-9-enoic acid) is a specific isomer of nitrated oleic acid
Drug: pravastatin — It is statin medicine used to lower cholesterol and triglycerides in the blood.
  Other Names: Pravachol®
Drug: Vytorin® (combination of simvastatin and ezetimibe) — It lowers bad cholesterol in the blood, and raises good cholesterol

SUMMARY:
This is an exploratory study in a small, well controlled group of healthy subjects to explore the effect of CXA-10 on pravastatin and Vytorin® (combination of simvastatin and ezetimibe).

DETAILED DESCRIPTION:
This is an exploratory study in a small, well controlled group of healthy subjects to explore the effect of CXA-10 on pravastatin and Vytorin® (combination of simvastatin and ezetimibe).

The overall design of the trial is to administer drugs that are metabolized through these transporters to quantify the impact CXA-10 may have on the exposure of these drugs.

The study will also examine the 24-h urine total creatinine excretion prior to and following administration of CXA-10 to examine the effects of CXA-10, if any, either directly on creatinine transporters or through enhanced creatinine production.

To reduce the potential variability in drug exposure levels, the study population will only include male subjects between 19 to 25 years of age.

ELIGIBILITY:
Inclusion Criteria:

* In good general health as determined by a thorough medical history and physical examination, ECG, vital signs, and clinical laboratory evaluation. Results of clinical laboratory tests must be without clinically significant abnormalities for this population and may exceed the limits of the reference ranges, including hematology, clinical chemistry and urinalysis except as noted below.
* Resting HR greater than or equal to 45 beats per minute (BPM) after 5 minute rest at screening.
* QTcF interval must be less than or equal to 430msec at screening and pre-dose.

Exclusion Criteria:

* Any clinically relevant abnormality for this population identified on the screening history, physical or laboratory examinations, or any other medical condition or circumstance making the volunteer unsuitable for participation in the study.
* Any clinical history of cardiovascular events, arrhythmias, fainting, palpitations, personal or family history of congenital prolonged QT syndromes or sudden unexpected death due to a cardiac reason.
* Treatment with any prescription or non-prescription drugs (including vitamins, herbal and dietary supplements) within 7 days or 5 half-lives, whichever is longer, prior to dosing and until collection of the final PK sample.
* History of smoking, including e-cigarettes, or use of nicotine-containing products within 1 month of screening.
* Subjects with any other clinically relevant ECG parameter abnormality (e.g., PR interval, QRS deviation) or any clinically significant ECG abnormality will be excluded from the study.

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blok, MD, Principal Investigator — Jasper Clinic, Michigan
Locations (1):
- Jasper Clinical Research & Development, Inc., Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No